CLINICAL TRIAL: NCT05711342
Title: The Added Value of an Internet-based Intervention for Treatment of Aggression in Forensic Psychiatric Outpatients: A Multicentre, Randomized Controlled Trial
Brief Title: The Added Value of an Internet-based Intervention for Treatment of Forensic Psychiatric Outpatients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Twente (Other)
Collaborators: Transfore (Unknown); Kairos (Unknown); GGZ Noord-Holland-Noord (Other); De Woenselse Poort (Unknown); Kwaliteit Forensische Zorg (KFZ) (Unknown)
Responsible Party: Principal Investigator, Hanneke Kip, Principal Investigator, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80846.091.22
Record Dates: First submitted 2022-06-17; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Aggression; Psychosocial Problem; Forensic Psychiatry; Internet-based Intervention
MeSH Terms: conditions — Aggression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) with a control condition that receives treatment as usual in forensic outpatient clinics, and an experimental condition that receives treatment as ususal plus the 10-week internet-based intervention 'Aggression'.
Masking Description: Because an internet-based intervention is used, patients, therapists and researchers cannot be blinded to the condition to which the participant is allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): In this control condition, participants receive in-person aggression treatment as usual (TAU). No changes to the way treatment is provided as usual are made. In general, this refers to any form of psychotherapy that is delivered by a licenced psychologist to a patient in a one-on-one setting. The main focus of treatment as usual should lie on aggression regulation. Additionally, patients should receive individual, one-on-one treatment and should not participate in group treatment of aggression during data collection.
  Interventions: Behavioral: Treatment as usual
- Treatment as usual (TAU) +Internet-based intervention Aggression (Experimental): In the experimental condition, participants receive TAU, and additionally work on the 10-week internet-based intervention 'Aggression', on which they can work in their own time, i.e. outside of treatment sessions. Consequenlty, the intervention is used in a blended way. The intervention is focused on three main objectives: (1) increasing the motivation to change, (2) acquiring skills for dealing with conflict, and (3) breaking the cycle of aggression by providing knowledge on situational, emotional, cognitive and physical triggers. The module consists of 10 lessons:
  Interventions: Behavioral: Aggression; Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Aggression — The intervention consists of 10 lessons:
  1. Motivation - where are you now?
  2. Where do you want to go?
  3. Circle of aggression.
  4. Thoughts.
  5. Emotions.
  6. Bodily sensations.
  7. Techniques for self-control.
  8. Asking for help.
  9. Assertiveness.
  10. Relapse-prevention. Each lesson consists of multiple components, i.e. written text, assignments and videos with therapists and/or experts by experience. After each lesson, the therapist sends written feedback on the assignments to the patient. Because 'Aggression' is a blended intervention, each lesson is briefly discussed in an in-person treatment session. Generally, participants work on one lesson per week.
  Other Names: Minddistrict
  Arms: Treatment as usual (TAU) +Internet-based intervention Aggression
Behavioral: Treatment as usual — In-person aggression treatment as usual (TAU), as delivered by the organization. This refers to any form of psychotherapy that is delivered by a licenced psychologist to a patient. The main focus of treatment as usual should lie on aggression regulation.

SUMMARY:
Even though internet-based interventions have been used in treatment of forensic psychiatric outpatients for over ten years, no robust research into their effectiveness has taken place. Multiple potential benefits and barriers have been observed in clinical practice, such as the possibility to increase a patient's treatment readiness, self-efficacy and thus reduce undesired behaviour such as reactive aggression. However, therapists indicate that these interventions do not seem to work for all forensic psychiatric patients, and that uptake is generally quite low. There is an urgent need to evaluate if and how these internet-based interventions are of added value for treatment of forensic psychiatric outpatients.

The main goal of this study is to investigate whether the addition of the existing internet-based intervention 'Aggression' to treatment as usual of forensic psychiatric outpatients leads to better treatment outcomes than treatment as usual that is delivered solely in-person.

This study uses a multicentre mixed methods randomized controlled trial (RCT) design, with four participating Dutch forensic psychiatric outpatient care organizations. Patients are included if they receive outpatient treatment for aggression regulation problems and will be randomized into an experimental condition, in which the internet-based intervention is added to treatment as usual (TAU), or a control condition, with only TAU. Participants are assessed four times: at baseline (T0), halfway during the 10-week intervention (T1), after completing the intervention (T2), and after three months (T3). Primary outcome measures are regulatory emotional self-efficacy, treatment readiness, and aggression, assessed via validated self-report questionnaires. Secondary outcome measures are the number of in-person treatment sessions during the data collection, and dynamic risk factors. Adherence to and engagement will be studied as potential predictors for effectiveness via respectively log data and a self-report questionnaire. Perceived benefits, barriers and points of improvement will be identified via qualitative interviews with participating patients and therapists.

This will be the first experimental study to investigate an internet-based intervention in a forensic psychiatric outpatient sample. By using a mixed-methods design and by adding adherence and engagement as potential predictors, this study can not only answer questions about if, but also why and for whom this intervention works. Consequently, this study will answer an important question from clinical practice: are these types of interventions - which have been used in practice for over ten years - actually of added value for treatment?

DETAILED DESCRIPTION:
Rationale: While internet-based interventions have been used for over ten years in Dutch forensic psychiatric outpatient care, no thorough evaluation study has been conducted yet. Studies on internet-based interventions in other mental healthcare sectors show promising results: they can increase the quality and efficiency of care. However, it is not clear if, why and for whom these interventions work in forensic mental healthcare. It is especially important to study whether these interventions are of added value for this complex patient population, known for its low treatment motivation, co-morbidity and low literacy levels.

Objective: The primary objective of this study is to investigate whether the addition of the internet-based intervention 'Aggression' to forensic psychiatric outpatient treatment as usual (TAU) results in better treatment outcomes in terms of self-reported regulatory emotional self-efficacy, treatment readiness, and aggression. Additionally, it is investigated whether the experimental group requires fewer treatment sessions and improves more on dynamic risk factors. Furthermore, to gain more insight into for whom these interventions work, it is investigated whether engagement with the internet-based intervention predicts adherence and effectiveness. Finally, this study aims to explore reasons for the (in)effectiveness of the intervention according to patients and therapists.

Study design: To investigate if the use of internet-based interventions is of added value for treatment of forensic psychiatric outpatients, a multicenter, non-blinded, parallel groups, randomized controlled trial design is used. Patients fill out three short self-report questionnaires four times: at baseline, mid-treatment (+6 weeks), post-treatment (+14 weeks) and at follow-up (+26 weeks). Semi-structured interviews with a randomly selected sample of 20 patients from the experimental condition and with all participating therapists are conducted to explain the results of the RCT.

Study population: The target group of this study consists of forensic psychiatric outpatients, treated in four Dutch organizations for aggression regulation problems.

Intervention (if applicable): This study investigates the existing internet-based intervention Aggression, which was introduced in forensic mental healthcare over ten years ago. However, as is the case with other internet-based interventions, uptake in practice remains relatively low. 'Aggression' is used as an addition to treatment as usual, and thus does not replace any part of treatment in this study. The intervention is earlier developed by the CE-certified company Minddistrict. The last couple of months the intervention has been cosmetically adjusted in close cooperation with therapists, patients and other stakeholders so that it fits the current design and lay-out of Minddistrict. The goals of this intervention are to (1) increasing the motivation to change, (2) acquiring skills for dealing with conflict, and (3) breaking the cycle of aggression by providing knowledge on situational, emotional, cognitive and physical triggers. It contains ten lessons, each containing written texts, videos and audio files, and short written assignments on which the therapist can give feedback.

Main study parameters/endpoints: All participants fill out three validated, short self-report questionnaires on self-efficacy, treatment readiness and aggression at four points during the study. Participants in the experimental conditions also fill out an engagement questionnaire during the use of the intervention. Dynamic risk factors are assessed via a risk assessment instrument that is already used as a standard part of treatment according to Dutch guidelines and the number of treatment sessions are retrieved from existing systems. The patient and therapist perspective is take in into account by means of semi-structured interviews.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since participants only have to fill out short questionnaires, participating in this study is not viewed as a major burden. Furthermore, interventions of Minddistrict have been used for over ten years in mental healthcare, during which no risks or adverse events have been observed. Because not all forensic psychiatric patients receive internet-based interventions as part of their standard care and because these interventions are not yet evaluated and are thus not evidence-based, participants in the control condition are not deprived of effective treatment. During the entire study, experienced therapists monitor the patient's progress. Finally, multiple precautions are taken to ensure that patients are aware that the decision to participate does not have any effect on their treatment progress. Consequently, the burdens and risks associated with this study are low or even non-existent.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. The patient is 18 years or older
2. The patient is treated at an outpatient clinic
3. The patient receives one-on-one treatment
4. During the intake, improvement of aggression regulation has been selected as one of the treatment objectives
5. The patient indicates that they are able to read and write simple texts
6. The therapist responsible for treatment of the patient indicates that participating will not result in any harm for the patient
7. The patient voluntarily consents to participation

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. The patient has a current psychosis
2. The patient resides in any type of psychiatric inpatient clinic - this can be a forensic, but also another type of clinic
3. The patient receives group treatment focused on aggression regulation (specifically: AR [aggressieregulatie] op maat)
4. The patient is analphabetic, i.e. being unable to read and write
5. The responsible therapists identifies any other valid reason for exclusion

As can be seen in the in- and exclusion criteria, the responsible therapist is actively involved in determining whether participating in the study is safe and possible for the patient. This will first be discussed during the MDO. If, after several treatment sessions, the therapist identifies any reasons for exclusion, this will be communicated to the researcher and the patient will not be invited to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Aggression | Change in aggression will be measured by assessing it on four time points before, throughout and after the use of the intervention: Assessed on T0 (Week 0), T1 (Week 6), T2 (Week 14), and T3 (Week 26)
  Change on self-reported aggression is assessed by means of the Dutch version of the much-used and validated Aggression Questionnaire (Aangepaste Versie van de Agressie Vragenlijst; AVL-AV). The 12 items of the questionnaire are divided into four subscales: physical aggression, verbal aggression, anger, and hostility. Items are scored on a 5-point Likert scale (min. total score = 12, max. total score = 60, higher scores indicate higher aggression levels).
Regulatory emotional self-efficacy | Change in regulatory emotional self-efficacy will be measured by assessing it on four time points before, throughout and after the use of the intervention: Assessed on T0 (Week 0), T1 (Week 6), T2 (Week 14), and T3 (Week 26)
  Change on regulatory emotional self-efficacy is measured by means of the validated, 12-item Regulatory Emotional Self-efficacy (RESE) scale. The RESE scale assesses self-efficacy in managing negative emotions (8 items) and in expressing positive emotions (4 items). Items are assessed via a 5-point Likert scale (min. total score = 12, max. total score = 60, higher scores indicate more regularoy emotional self-efficacy). Negative emotional self-efficacy refers to the perceived "capability to ameliorate negative emotional states once they are aroused in response to adversity or frustrating events and to avoid being overcome by emotions such as anger, irritation, despondency, and discouragement". Positive self-efficacy is defined as the perceived capability "to experience and to allow oneself to express positive emotions such as joy, enthusiasm and pride in response to success or pleasant events".
Treatment readiness | Change in treatment readiness will be measured by assessing it on four time points before, throughout and after the use of the intervention: Assessed on T0 (Week 0), T1 (Week 6), T2 (Week 14), and T3 (Week 26)
  Treatment readiness refers to the presence of factors that contribute to engagement with treatment and therapeutic change. Change in treatment readiness is assessed by the Dutch version of the Corrections Victoria Treatment Readiness Questionnaire (CVTRQ): a validated self-reported questionnaire. The total scale consists of 20 items and uses a 5-point Likert scale (min. total score = 20, max total score = 100, higher scores indicate higher treatment readiness).
  The CVTRQ is divided into four subscales. The subscale Attitude and Motivation (AM) measures attitudes and beliefs about treatment programs and the desire to change. The scale Emotional reactions (ER) measures emotional responses to the individual's offending behaviour. Offending beliefs (OB) refers to beliefs about personal responsibility for offending behaviour. The subscale Efficacy (EF) measures perceived ability to participate in treatment programs.

SECONDARY OUTCOMES:
Risk assessment - dynamic risk factors | Assessed on T0 (Week 0) and T3 (Week 26)
  In treatment of all forensic psychiatric patients, risk assessment has to be conducted by means of evidence-based risk assessment instruments. In forensic psychiatric outpatient care, the Dutch standard is the Forensisch Ambulante Risico Evaluatie (FARE), version 2 [36]. The FARE is not only used to estimate the risk on recidivism, but also to monitor changes in dynamic risk factors and risk of recidivism during treatment.

OTHER OUTCOMES:
Engagement | Assessed only in the experimental group (TAU + Aggression) on T0 (week 0), T1 (week 6) and T2 (week 14).
  Engagement is a non-specific factor that can be used to predict effectiveness of and adherence to internet-based interventions. Engagement refers to the extent to which someone is involved or occupied with something, and is often related to a positive outcome, such as effectiveness.this study, engagement is measured with the TWente Engagement with Ehealth and Technologies Scale (TWEETS). The scale employs a definition of engagement that incorporates behaviour, cognition, and affect and comprises of 9 items, all scored on a 5-point Likert scale (min. total score = 9, max. total score = 45, higher scores mean more engagement).

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Kairos, Nijmegen, Gelderland
  - De Woenselse Poort, Eindhoven, North Brabant
  - GGZ Noord-Holland-Noord, Heiloo, North Holland
  - Transfore, Deventer, Overijssel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to site of grant provider on the project — https://kfz.nl/projecten/de-effectiviteitspuzzel-van-ehealth

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05711342/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT05711342/ICF_001.pdf